CLINICAL TRIAL: NCT04831047
Title: The Effect of Upneeq (Oxymetazoline Hydrochloride 0.1%) on Palpebral Fissure Height, Eye Redness, and Patient-reported Eye Appearance
Brief Title: The Effect of Upneeq (Oxymetazoline Hydrochloride 0.1%) on Eyelid Position, Eye Redness, and Eye Appearance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Wendy Lee, Associate Professor of Ophthalmology and Dermatology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210199
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Ptosis, Eyelid; Conjunctiva Inflamed; Eye Manifestations
MeSH Terms: conditions — Blepharoptosis; Conjunctivitis; Eye Manifestations | interventions — Oxymetazoline; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Upneeq Group (Experimental): Participants in this group will receive a one-time dosing of oxymetazoline hydrochloride 0.1% (1 drop applied to ocular surface of each eye of patients in the treatment group)
  Interventions: Drug: Oxymetazoline hydrochloride 0.1% ophthalmic solution
- Control Group (Sham Comparator): Participants in this group will receive a one-time dosing of balanced saline solution (1 drop applied to ocular surface of each eye of patients in the control group)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxymetazoline hydrochloride 0.1% ophthalmic solution — One drop of Upneeq (Oxymetazoline hydrochloride 0.1% ophthalmic solution) will be applied to the ocular surface of each eye.
  Other Names: Upneeq
  Arms: Upneeq Group
Drug: Placebo — One drop of placebo (balanced saline solution) will be applied to the ocular surface of each eye.
  Other Names: Balanced saline solution
  Arms: Control Group

SUMMARY:
The purpose of the research is to see if Upneeq ( oxymetazoline 0.1% ophthalmic solution) has an effect on eyelid position, eye redness, or patient-perceived appearance of the eyes.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and above able to provide informed consent to participate
* Subject with stable ocular health, defined as no ocular conditions requiring ongoing topical therapy or recent surgical intervention

Exclusion Criteria:

* Adults unable to consent
* Individuals less than 18 years of age
* Prisoners
* Pregnant women.
* Known contradictions or sensitivities to study medication (oxymetazoline)
* Ocular surgery within the past 3 months or refractive surgery within the past six months
* Grossly abnormal lid margins, anatomical abnormalities, previous eyelid or orbital surgery
* Variable ptosis or eyelid position (e.g., myasthenia gravis, thyroid eye disease, or blepharospasm)
* Any ocular or systemic condition that, in the opinion of the investigator, would confound study data, interfere with the subject's study participation, or affected the subject's safety or trial parameters
* Presence of an active ocular infection
* Prior (within 5 days of beginning study treatment) use of eye whiteners (eg, vasoconstrictors), decongestants, antihistamines (including over the counter and herbal topical ophthalmic medications), phenylephrine dilating drops, any other topical ophthalmic agents
* Inability to sit comfortably for 15 - 30 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy W. Lee, MD, Principal Investigator — University of Miami Bascom Palmer Eye Institute
Locations (1):
- University of Miami Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shoji MK, Markatia Z, Ameli K, Bayaraa M, Clauss KD, Ugradar S, Lee WW. The effects of topical oxymetazoline on eyelid position, eye redness, and patient-reported eye appearance: A randomized controlled trial. J Plast Reconstr Aesthet Surg. 2023 May;80:66-74. doi: 10.1016/j.bjps.2023.02.006. Epub 2023 Feb 9. PMID 36996503

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Upneeq Group | Control Group
Started | 57 | 57
Completed | 57 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Upneeq Group | Control Group | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (12.7) | 31.3 (10.1) | 33.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 18 | 19 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 26 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 40 | 28 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Palpebral Fissure [Mean (Standard Deviation); unit: mm] | 10.1 (1.5) | 10.5 (1.7) | 10.3 (1.6)
Eye Redness [Mean (Standard Deviation); unit: units on a scale] — Scoring of ocular redness from clinical photographs will be performed by investigators on a 10 - 100 unit scale as compared to standardized reference photographs per the Validated Bulbar Redness grading scale (10 = minimal redness, 100 = very red) before and after drop instillation. Higher score indicates more redness.
  units on a scale | 13.2 (4.7) | 12.1 (4.1) | 12.6 (4.4)
FACE-Q Eye Appearance [Mean (Standard Deviation); unit: units on a scale] — Population: One patient did not complete FACE-Q survey in control group
  units on a scale
    number analyzed (Participants) | 57 | 56 | 113
    (all) | 21.2 (4.7) | 22.7 (4.1) | 21.9 (4.4)
FACE-Q Upper Eyelid Appearance [Mean (Standard Deviation); unit: units on a scale] — Population: One patient did not complete FACE-Q survey in control group
  units on a scale
    number analyzed (Participants) | 57 | 56 | 113
    (all) | 23.4 (5.8) | 24.3 (4.7) | 23.8 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Palpebral Fissure Height
Description: Palpebral fissure height will be calculated from the sum of marginal reflex distance 1 and 2 measured from the photograph by Ipad software and recorded by investigators before and after drop instillation.
Time Frame: Baseline, Day 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Upneeq Group | Control Group
Number analyzed (Participants) | 57 | 57
mm | 1.1 (1.1) | -0.4 (0.8)

2. Secondary Outcome: Change in Eye Redness as Measured by the Validated Bulbar Redness Grading Scale
Description: Scoring of ocular redness from clinical photographs will be performed by investigators on a 10 - 100 unit scale as compared to standardized reference photographs per the Validated Bulbar Redness grading scale (10 = minimal redness, 100 = very red) before and after drop instillation. Higher score indicates more redness.
Time Frame: Baseline, Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Upneeq Group | Control Group
Number analyzed (Participants) | 57 | 57
units on a scale | -2.6 (4.4) | -0.5 (2.3)

3. Secondary Outcome: Change in Patient-reported Eye Appearance - FACE-Q Eye Appearance
Description: Change in patient-reported eye appearance will be assessed by patient completion of the FACE-Q Eye Module Survey assessing overall eye appearance with a sum score of 7 (worst) to 28 (best) at baseline and after drop administration. Higher score indicates a higher level of satisfaction with eye appearance.
Time Frame: Baseline, Day 1
Population: One control patient declined completion of FACE-Q survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upneeq Group | Control Group
Number analyzed (Participants) | 57 | 56
score on a scale | 4.2 (5.4) | 0.8 (3.8)

4. Secondary Outcome: Change in Patient-reported Eye Appearance - FACE-Q Upper Eyelid Appearance
Description: Change in patient-reported upper eyelid appearance will be assessed by patient completion of the FACE-Q Eye Module Survey assessing overall upper eyelid appearance with a sum score of 7 (worst) to 28 (best) at baseline and after drop administration. Higher score indicates a higher level of satisfaction with upper eyelid appearance.
Time Frame: Baseline, Day 1
Population: One control patient declined completion of FACE-Q survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upneeq Group | Control Group
Number analyzed (Participants) | 57 | 56
score on a scale | 0.9 (4.9) | -0.5 (4.8)

ADVERSE EVENTS:
Time Frame: 1 day: this study was a single time-instillation of a topical temporary medication
Arm/Group | Upneeq Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 7/57 | 5/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upneeq Group (N=57) | Control Group (N=57)
Dry eye (Eye disorders) | 3 (3) | 2 (2)
Headache (General disorders) | 2 (2) | 1 (1)
Eyelid heaviness (Eye disorders) | 3 (3) | 0 (0)
Light Sensitivity (Eye disorders) | 1 (1) | 0 (0)
Temporary Blurry Vision (Eye disorders) | 0 (0) | 1 (1) — Lasted 10 minutes after drop instillation
Dizziness (General disorders) | 0 (0) | 1 (1) — Self-resolving dizziness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT04831047/Prot_SAP_000.pdf